CLINICAL TRIAL: NCT06513923
Title: Comparative Study of Remimazolam, Remimazolam Plus Flumazenil vs Propofol Anesthesia on Emergence Time in Elderly Patients Undergoing Hip Replacement: A Randomized, Double Blinded Controlled Study
Brief Title: Comparison of Remimazolam and Propofol on Emergence in Elderly Orthopedic Patients Under General Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Ru-Ping Dai, professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LYG2023002
Record Dates: First submitted 2024-07-05; First posted 2024-07-22 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Hip Fracture
MeSH Terms: conditions — Hip Fractures | interventions — remimazolam; Flumazenil; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remimazolam group (Experimental): Patients will receive remimazolam for induction and maintenance of anesthesia.
  Interventions: Drug: Remimazolam
- Remimazolam + Flumazenil group (Experimental): Patients will receive remimazolam for induction and maintenance, followed by flumazenil to reverse its effects.
  Interventions: Drug: Remimazolam; Drug: Flumazenil
- Propofol group (Experimental): Patients will receive propofol for induction and maintenance of anesthesia.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — In Remimazolam group, the induction dose of remimazolam is 0.3 mg/kg based on previous studies, the maintenance of anesthesia is 0.3-0.7 mg/kg/hr.
  Arms: Remimazolam + Flumazenil group; Remimazolam group
Drug: Flumazenil — Immediately after the cessation of remimazolam infusion in PACU(PACU, Postanesthesia care unit), the nurses who are blind to the anesthesia management were asked to administer the flumazenil.
  Arms: Remimazolam + Flumazenil group
Drug: Propofol — For propofol group, the induction of propofol is 1.5-2.0 mg/kg, followed by the maintenance of propofol infusion with 6-8 mg/kg/hr throughout the surgical procedure.
  Arms: Propofol group

SUMMARY:
Purpose: This study aims to compare the emergence time among three anesthesia regimens: remimazolam, remimazolam with flumazenil, and propofol in elderly patients undergoing hip replacement surgery.

Background: Previous studies have shown that flumazenil accelerates emergence time when used with remimazolam. Remimazolam and propofol have comparable emergence times, although remimazolam can be up to 5 minutes longer than propofol.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (≥65 years old).
* Scheduled for elective hip replacement surgery.
* ASA (ASA, American Society of Anesthesiologists) physical status I-III.
* Able to provide informed consent.

Exclusion Criteria:

* Known hypersensitivity to remimazolam, flumazenil, or propofol.
* Severe hepatic or renal impairment.
* History of benzodiazepine or alcohol abuse.
* Cognitive impairment that may interfere with the ability to provide consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 136 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Time to Emergence | Within one day of surgery
  Defined as the time from discontinuation of the anesthetic agent to the time the patient opens their eyes on verbal command.

SECONDARY OUTCOMES:
Hemodynamic Parameters | During operation
  Blood pressure measured at various time points including diastolic and systolic blood pressure.
Hemodynamic Parameters | During operation
  Heart rate measured at various time points.
Post-Operative Recovery | Within one day of surgery
  Assessed using the Modified Aldrete Score.The modified Aldrete score is measured by evaluating five criteria, including the individual's activity level, respiration, circulation, consciousness, and oxygen saturation. A score of "0", "1", or "2" is given for each category, two representing the ideal condition.Given the five parameters, individuals can have a total score from zero to ten. A score lower than nine typically means the individual's status is suboptimal.
Adverse Events | Within one day of surgery
  Incidence and severity of adverse events related to anesthesia(injection pain, post-induction hypotension, bradycardia and body movement, postoperative nausea and vomiting, intraoperative awareness and delirium, sedation rescue and re-sedation).

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Ping MD Dai, PhD, Principal Investigator — Central South University
Locations (2):
- China (2):
  - Department of Anesthesiology, The Second Xiangya Hospital, Changsha, Hunan
  - The Second Xiangya Hospital, Changsha, Hunan